CLINICAL TRIAL: NCT00336765
Title: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of XL647 Administered Orally Daily to Subjects With Solid Tumors
Brief Title: Study of XL647 Administered Orally Daily to Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL647-002
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Cancer
Keywords: solid tumors
MeSH Terms: conditions — Neoplasms | interventions — XL647

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL647 — Tablets supplied in 50-mg strength administered orally daily
  Other Names: KD019

SUMMARY:
The purpose of this study is to assess the safety and tolerability of the multiple receptor tyrosine kinase (RTK) inhibitor (including EGFR, VEGFR2, ErbB2, and EphB4) XL647 when given orally daily to adults with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically confirmed malignancy that is metastatic or unresectable
* Subject has disease that is assessable by tumor marker, physical, or radiologic means
* Subject is at least 18 years old
* Subject has an ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
* Subject has a life expectancy ≥ 3 months
* Subject has normal organ and marrow function
* Subject gives written informed consent
* Subject must use an accepted method of contraception during the study
* Female subjects of childbearing potential must have a negative pregnancy test

Exclusion Criteria:

* Subject has received anticancer treatment within 30 days of first dose of XL647
* Subject has received another investigational agent within 30 days of first dose of XL647
* Subject has known brain metastases
* Subject has corrected QT interval (QTc) of > 0.45 seconds
* Subject is currently receiving anticoagulation therapy with warfarin
* Subject has uncontrolled intercurrent illness
* Subject is pregnant or breastfeeding
* Subject has known HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Evaluate safety, tolerability, and maximum tolerated dose of XL647 | Inclusion until 30 days post last treatment

SECONDARY OUTCOMES:
Characterize pharmacokinetics and pharmacodynamic effects of XL647 | At various time points from pre-dosing until post dosing
Evaluate preliminary tumor response | Inclusion until disease progression

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University Medical Center, Stanford, California
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Background] Das M, Padda SK, Frymoyer A, Molina J, Adjei A, Lensing JL, Miles D, Sikic BI, Wakelee HA. A safety, tolerability, and pharmacokinetic analysis of two phase I studies of multitargeted small molecule tyrosine kinase inhibitor XL647 with an intermittent and continuous dosing schedule in patients with advanced solid malignancies. Cancer Chemother Pharmacol. 2018 Sep;82(3):541-550. doi: 10.1007/s00280-018-3646-0. Epub 2018 Jul 20. PMID 30030583